CLINICAL TRIAL: NCT01119508
Title: Phase II Study of Ipilimumab Plus Temozolomide in Patients With Metastatic Melanoma
Brief Title: Ipilimumab + Temozolomide in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0408; NCI-2011-00565 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Melanoma
Keywords: Advanced; Inoperable; Melanoma; Ipilimumab; MDX010; BMS-734016; Temozolomide; Temodar; TMZ; skin; mucosal
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab + Temozolomide (Experimental): Induction: Ipilimumab 10 mg/kg IV over 90 minutes Day 1 + Temozolomide 200 mg/m2 PO on Days 1 - 4, every 3 weeks for 4 courses over 3 months.
  Interventions: Drug: Ipilimumab; Drug: Temozolomide

INTERVENTIONS:
Drug: Ipilimumab — Induction Phase: 10 mg/kg by vein (IV) over approximately 90 minutes on Day 1 only repeated every 3 weeks until 4 courses of therapy are given over 3 months. For the Maintenance Phase, dose repeated every 12 weeks.
  Other Names: BMS-734016; MDX010
Drug: Temozolomide — Induction Phase, 200 mg/m^2 by mouth (PO) on Days 1 to 4, repeated every 3 weeks until 4 courses of therapy are given over 3 months. For the Maintenance Phase, dose delivered on Days 1 to 5, repeated every 4 weeks.
  Other Names: Temodar

SUMMARY:
The goal of this clinical research study is to learn if combining ipilimumab and temozolomide can help to control metastatic melanoma. The safety of this drug combination will be studied. Researchers would also like to study how this therapy affects the levels of certain chemicals in the blood that are related to your immune system.

DETAILED DESCRIPTION:
The ability to control melanoma depends on how well your immune system recognizes and then attacks cancer cells. Researchers want to use ipilimumab to try to trigger your immune system response, while temozolomide is designed to damage the cancer cells themselves.

Study Drugs:

Ipilimumab is designed to block the activity of cells that lower the immune system's ability to fight cancer. Blocking these cells may help the body's immune system fight the cancer cells better.

Temozolomide is designed to stop cancer cells from making new DNA (the genetic material of cells). If they cannot make DNA, then they cannot divide into new cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will begin to receive treatment with ipilimumab plus temozolomide. You will have an intravenous (IV) catheter placed into a large vein for the Ipilimumab.

There are 2 phases of study drug treatment: Induction and Maintenance.

During the Induction Phase, you will receive ipilimumab by vein over 90 minutes on Day 1 of each 3-week Induction "course." You will take temozolomide by mouth in tablet form on Days 1-4 of each course. You will receive up to 4 courses of Induction therapy.

During the Maintenance Phase, you will receive ipilimumab by vein over 90 minutes on Day 1 every 12 weeks. You will also take temozolomide by mouth for 5 days in a row, every 4 weeks.

You may take the Temozolomide dose within 48 hours of receiving the Ipilimumab dose on Day 1 of both the Induction and the Maintenance Phase.

You will see your doctor before each new course (every 3 weeks) during the Induction Phase, and once every 4 weeks during the Maintenance Phase. All treatments will be given in the outpatient clinic. You will be given anti-nausea medication to decrease the risk of nausea and vomiting, as needed.

Study Tests:

Before Each Course:

(Every 3 weeks during Induction, and every 4 weeks during Maintenance)

* Blood (about 1 teaspoon) will be drawn for routine tests and tests of your liver and kidney function.
* You will be asked about any medication you are taking and any side effects you are experiencing.
* Women who are able to become pregnant will have a blood (about 1 teaspoon) or urine pregnancy test.
* Your performance status will be recorded.
* Your vital signs will be measured on Day 1.

Every week, blood (about 1 teaspoon) will be drawn for routine tests.

At the end of each course, any tumor that can be felt with the hands will be measured during physical exam to see if it is shrinking.

Every 2 courses (+/- 7 days), you will have a chest x-ray and CT or MRI scans performed to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

If you stop receiving the study drugs for any reason, you will have an End-of-Treatment Visit.

End-of-Treatment Visit:

Within 14 days after you stop study treatment, you will come into the clinic for the End-of-Treatment Visit. At this visit, the following tests will be performed:

* You will have a physical exam, including a measurement of your vital signs and weight.
* You will be asked about any other medications you are taking or any side effects you are experiencing.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* Your may have a CT or MRI scan performed to check for side effects.

Every 2 months for up to 3 years, you will also be contacted by telephone or during a clinic visit to see how you are doing.

This is an investigational study. At this time, temozolomide is FDA approved and commercially available for the treatment of primary brain cancer. However, the use of temozolomide in treating metastatic melanoma is considered investigational. At this time, ipilimumab is being used in research only. The use of these drugs together is also considered investigational.

Up to 64 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced/inoperable metastatic melanoma of skin or mucosal origin are eligible, provided they fulfill the following conditions:
2. They are 18 years old to 75 years old with measurable (at least 1 cm) metastatic disease.
3. They have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Must be at least 21 days since surgery, radiation therapy and 6 weeks after immunotherapy with regimens including vaccine, interferon, IL-2 etc. and fully recovered from adverse effects of these therapies.
5. Must agree not use vaccines for the treatment of cancer or prevention of disease unless indicated as a component of the protocol regimen (including those for common medical conditions) for up to one month pre and post dosing with ipilimumab.
6. Required values for initial laboratory tests: white blood cell count (WBC): 2000/uL or greater, absolute neutrophil count (ANC): 1000/uL or greater, Platelets: 100 x 103/uL or greater, Hemoglobin: 9 g/dL or greater, Creatinine: </=1.5 mg/dL, AST and ALT: </= 2.5 x upper limit of normal (ULN) for subjects without liver metastasis or, </= 5 X upper limit of normal (UNL) for liver metastases, Bilirubin: </= 1.5 mg/dL, LDH </= 2 X upper limit of normal (UNL).
7. They have no significant intercurrent illness such as a serious infection which requires intravenous antibiotics. No active or chronic infection with HIV, Hepatitis B, or Hepatitis C. No significant psychiatric illness, which includes any life threatening psychiatric illness that has not been adequately controlled despite intervention (with or without medication) despite 6 months of therapy. They should have no GI tract metastasis or bleeding, no autoimmune disease.
8. They have not been previously exposed to any cytotoxic drugs, targeted therapies or anti CTLA 4 drugs for metastatic melanoma. Patients that received interferon for melanoma in the adjuvant setting are eligible. Prior radiation therapy for metastatic melanoma is permitted provided the patient has unirradiated metastatic sites for response evaluation and any toxicity has returned to baseline.
9. Patients with brain metastases who have been treated with craniotomy and resection or stereotactic radiosurgery of all symptomatic brain metastases are eligible provided they are 4 weeks from the procedures, MRI/CT of the brain performed within 3 weeks from registration fails to show new metastases and they are off of steroids for at least 2 weeks. Patients previously treated with whole brain radiotherapy are eligible if they are without tumor progression in the brain at least 8 weeks from completion of radiotherapy and are asymptomatic. They should be off steroid therapy for at least 2 weeks.
10. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. In general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject.
11. (Continued 10) WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as: 1) Amenorrhea 12 consecutive months without another cause, or 2) For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level 35 milli-International unit (mIU)/mL.
12. (Continued 11) Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.
13. Men should use condoms while participating in this study.
14. must agree not to use vaccines for the treatment of cancer or prevention of disease unless indicated as a component of the protocol regimen (including those for common medical conditions) for up to one month pre and post dosing of ipilimumab.

Exclusion Criteria:

1. Patients with Uveal melanoma. Patients with skin or mucosal melanoma who are younger than 18 years or more than 75 years of age and those with an ECOG performance status of 2, 3 or 4, or patients without measurable metastases.
2. Patients with prior cytotoxic, targeted therapy or anti-CTLA 4 drugs for metastatic disease.
3. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function or serious cardiac arrhythmias requiring therapy. Borderline cases must be discussed with the PI.
4. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD). Pulmonary function test with the results forced expiratory volume at one second (FEV1) <65% or forced vital capacity (FVC) <65% of predicted. Borderline cases must be discussed with the PI.
5. Patients on corticosteroids or any other type of immunosuppressive agent (e.g., methotrexate, chloroquine, azathioprine, cyclophosphamide) at time of enrollment only.
6. Patients with history of second malignancies such as basal cell carcinoma, squamous cell carcinoma and carcinoma in situ of cervix are eligible for therapy. Patients with history of other types of cancers, are eligible provided that they have been free of recurrence from second malignancy for at least 3 years. Each case must be discussed with the PI prior to registration.
7. Patients with symptomatic uncontrolled brain metastasis that is associated with significant brain edema requiring steroid therapy. Patients will be evaluated by the principal investigator or his designee. Patients with spinal cord metastasis or meningeal carcinomatosis.
8. WOCBP who are unwilling or unable to use an acceptable contraceptive method to avoid pregnancy. Acceptable contraceptive methods are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna P. Patel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 26, 2010 to August 29, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Ipilimumab + Temozolomide: Induction: Ipilimumab 10 mg/kg intravenous (IV) over 90 minutes Day 1 repeated every 3 weeks until 4 courses of therapy are given over 3 months + Temozolomide 200 mg/m2 orally Days 1 to 4; both repeated every 3 weeks for 4 courses over 3 months. For Maintenance Phase, Ipilimumab repeated every 12 weeks, Temozolomide Days 1 to 5 repeated every 4 weeks.
Period: Overall Study
Arm/Group | Ipilimumab + Temozolomide
Started | 64
Received Four Induction Doses | 45
Received Fifth Consolidation Dose week12 | 32
Completed | 5
Not Completed | 59
Not completed — Adverse Event | 56
Not completed — Withdrawal by Subject | 2
Not completed — Died before tumor response evaluation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab + Temozolomide
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: 6-Month Progression-Free Survival (PFS) Rate
Description: 6-month progression free survival rate is defined as the number of participants without progression per RECIST 1.0 6 months after starting study treatment.
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Ipilimumab + Temozolomide
Number analyzed (Participants) | 64
participants | 29

ADVERSE EVENTS:
Time Frame: Adverse Events collected till 30 days after the last dose of drug, approximate total of 7 weeks for Induction and Maintenance periods.
Arm/Group | Ipilimumab + Temozolomide
All-Cause Mortality (participants affected / at risk) | 1/64
Serious Adverse Events (participants affected / at risk) | 59/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + Temozolomide (N=64)
Pruritis (Skin and subcutaneous tissue disorders) | 4
Skin rash (Skin and subcutaneous tissue disorders) | 7
Fatigue (General disorders) | 10
Nausea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Anorexia (Gastrointestinal disorders) | 1
Pain (General disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
ALT (high) (Metabolism and nutrition disorders) | 3
AST (high) (Metabolism and nutrition disorders) | 3
Alk Phos (high) (Metabolism and nutrition disorders) | 1
Total Bilirubin (high) (Metabolism and nutrition disorders) | 1
Magnesium (low) (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + Temozolomide (N=64)
Pruritis (Skin and subcutaneous tissue disorders) | 52
Skin rash (Skin and subcutaneous tissue disorders) | 46
Fatigue (General disorders) | 40
Nausea (Gastrointestinal disorders) | 48
Constipation (Gastrointestinal disorders) | 44
Diarrhea (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 33
Anorexia (Gastrointestinal disorders) | 32
Dry Skin (Skin and subcutaneous tissue disorders) | 33
Headache (Nervous system disorders) | 32
Pain (Musculoskeletal and connective tissue disorders) | 18
Fever (General disorders) | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Colitis (Gastrointestinal disorders) | 6
Anemia (Blood and lymphatic system disorders) | 42
Neutropenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Hyperglycemia (Metabolism and nutrition disorders) | 41
ALT (high) (Metabolism and nutrition disorders) | 26
AST (high) (Metabolism and nutrition disorders) | 24
Alk Phos (high) (Metabolism and nutrition disorders) | 15
Total Bilrubin (high) (Metabolism and nutrition disorders) | 9
Magnesium (low) (Metabolism and nutrition disorders) | 16
Creatinine (high) (Metabolism and nutrition disorders) | 16
Potassium (low) (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes